CLINICAL TRIAL: NCT06343129
Title: Effects of an Education Program Emphasizing a Whole-food, Plant-based Nutrition Program on Blood Pressure and Blood Potassium Levels in Subjects With Chronic Kidney Disease
Brief Title: Effects of a Whole-food, Plant-based Nutrition Program on BP and Potassium in Subjects With CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Rochester Lifestyle Medicine Institute (Unknown)
Responsible Party: Principal Investigator, Scott Liebman, Professor of Medicine, Division of Nephrology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3817
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Diseases
Keywords: Diet; Plant-based; Whole food; Hypertension; Hyperkalemia; Blood pressure; Potassium; Systolic blood pressure; Diastolic blood pressure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Hyperkalemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jumpstart Educational Program (Experimental): Jumpstart sessions on day 1, 2, 5, 8, 12, and 15. Tests at baseline and week 2 visit: blood pressure, height and weight measurements to calculate a body mass index, urine tests to assess antioxidant activity, quality of life questionnaire (~8 minutes to complete) about physical and mental symptoms, a 3-day food record to assess if participants are changing their diet over the course of the study, assessment of medication use.
  Tests performed at day 1, day 8, and day 15: A small blood draw [about 1 teaspoon] to check chemistry levels, cholesterol, and markers of inflammation. Laboratory tests are reviewed once available, and participant contacted by the study team either by telephone or My Chart regarding clinically significant results that require intervention. If potassium levels are higher than 5.2 Meq/L, the study team contacts the participant or their alternate contact directly. For the intervention group, this is in addition to the finger-stick blood collection.
  Interventions: Behavioral: Dietary education program
- Control group (No Intervention): Participants randomized to the control group continue to receive medical, dietary, and nutritional advice from their medical team as normal. The testing is the same testing as the intervention group and will be done at day 1, day 8, and day 15 of the study. They do not participate in the educational sessions during the study but will have the opportunity to participate in the program at no charge at the conclusion of the study.

INTERVENTIONS:
Behavioral: Dietary education program — Jumpstart educational program:
  https://www.rochesterlifestylemedicine.com/about-community-jumpstart/
  Other Names: Nutritional education program
  Arms: Jumpstart Educational Program

SUMMARY:
The purpose of this study is to determine if an educational program emphasizing a whole food plant based diet favorably impacts blood pressure while not significantly increasing blood potassium levels, by comparing a group of patients receiving the educational program with a control group of patients receiving no specific education.

DETAILED DESCRIPTION:
The primary objective of this study is to test the hypothesis that educating hypertensive chronic kidney disease (CKD) stage 3 and 4 patients on the benefit of a whole food plant based (WFPB) diet in the context of a 15-day educational program ("Jumpstart program") will lead to improved blood pressure control and will not increase rates of hyperkalemia.

Other objectives:

A) To test the effect of the Jumpstart program on degree of uptake on a WFPB diet via a 3 day food recall.

B) To test the effect of the Jumpstart program on other important outcomes in CKD in the following domains:

1. Body composition such as weight and body mass index (BMI).
2. Quality of life.
3. Laboratory tests including- serum levels of sodium, bicarbonate, chloride, Blood urea nitrogen, creatinine, calcium, phosphorus, magnesium, albumin, parathyroid hormone, fibroblast growth factor 23, lipids, C-reactive protein and erythrocyte sedimentation rate.

C) To test the effect of the Jumpstart program on quality of life in hypertensive CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Subjects with CKD 3 and 4 (as determined by an estimated glomerular filtration rate of ≥ 15 ml/min but < 60 ml/min for at least three months)
* Subjects with hypertension, defined as use of antihypertension medication:
* Lack of significant proteinuria ( subjects will have a 24 hour urine protein value of < 500 mg or a spot protein to creatinine ratio of < 0.5 or a microalbumin to creatinine ratio < 300) within previous 3 months.
* Fluent in English language
* Able and willing to comply with the testing schedule and the meeting schedule of the Jumpstart
* Able and willing to comply with dietary advice of whole-food plant based diet given during the educational session
* Able and willing to give informed consent
* Must have computer/internet access to participate in virtual Zoom educational sessions (intervention group only)

Exclusion Criteria:

* Kidney disease requiring immunosuppressive therapy
* Diabetes mellitus
* Pregnancy
* Life expectancy < 12 months
* History of solid organ transplant or anticipated solid organ transplant in next 2 months
* History of hyperkalemia: (two or more potassium levels ≥ 5.0 Meq/L or those requiring intervention for high potassium levels within the last six months)
* Subjects with malabsorptive syndromes
* Subjects with history of bariatric surgery or planned bariatric surgery in the next 2 months
* Subjects on warfarin
* Subjects with documented eating disorder at the time of consent
* Allergy or intolerance of a plant-based or plant-derived food (gluten, soy, etc.)
* Following a vegan diet in the six months prior to consent
* Major surgery within 60 days prior to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Mean change in systolic blood pressure | Baseline to day 15
  Unit of measurement - mm Hg
Mean change in diastolic blood pressure | Baseline to day 15
  Unit of measurement - mm Hg
Mean change in potassium levels | Baseline to day 15
  Unit of measurement - mEq/L
Proportion of participants developing hyperkalemia | Day 15
  Percentage

SECONDARY OUTCOMES:
Mean Change in energy/day | Baseline to day 15
  Unit of measurement - kcal/day. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in energy/kg of body mass | Baseline to day 15
  Unit of measurement - kcal/kg/day. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in total fat | Baseline to day 15
  Unit of measurement - grams. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in % calories from fat | Baseline to day 15
  Unit of measurement - Percentage. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in % calories from carbohydrates | Baseline to day 15
  Unit of measurement - Percentage. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in % calories from protein | Baseline to day 15
  Unit of measurement - Percentage. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in Animal protein | Baseline to day 15
  Unit of measurement - grams. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in Vegetable protein | Baseline to day 15
  Unit of measurement - grams. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in cholesterol | Baseline to day 15
  Unit of measurement - milligrams. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in Total dietary fiber | Baseline to day 15
  Unit of measurement - grams. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in Total fiber per 1000 kcal | Baseline to day 15
  Unit of measurement - Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in calcium | Baseline to day 15
  Unit of measurement - milligrams. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in phosphorous | Baseline to day 15
  Unit of measurement - milligrams. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in magnesium | Baseline to day 15
  Unit of measurement - milligrams. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in sodium | Baseline to day 15
  Unit of measurement - milligrams. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in potassium | Baseline to day 15
  Unit of measurement - milligrams. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in body mass | Baseline to day 15
  Unit of measurement - kilograms. Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in body mass index | Baseline to day 15
  Unit of measurement - kg/m². Subjects completed a 3-day food record prior to intervention and during Jumpstart (or equivalent time for controls). Participants were given a recording form, and verbal and written instructions to record relevant details for all foods and beverages consumed. Portion size was estimated, using food visual aids, or measured, using weight scales or volume measures. A research dietitian (NW) provided the food record instruction and reviewed the completed records with participants to increase the quality of the report. The food record data was then entered into the Nutrition Data System for Research (NSDR, Nutrition Coordinating Center, University of Minnesota, Twin Cities) for calculation of nutrient intake.
Mean change in sodium measured in blood | Baseline to day 15
  Unit of measurement - mEq/L
Mean change in chloride measured in blood | Baseline to day 15
  Unit of measurement - mEq/L
Mean change in bicarbonate measured in blood | Baseline to day 15
  Unit of measurement - mEq/L
Mean change in blood urea nitrogen (BUN) measured | Baseline to day 15
  Unit of measurement - mg/dl
Mean change in creatinine measured in blood | Baseline to day 15
  Unit of measurement - mg/dl
Mean change in glucose measured in blood | Baseline to day 15
  Unit of measurement - mg/dl
Mean change in calcium measured in blood | Baseline to day 15
  Unit of measurement - mg/dl
Mean change in phosphorous measured in blood | Baseline to day 15
  Unit of measurement - mg/dl
Mean change in parathyroid hormome (PTH) measured in blood | Baseline to day 15
  Unit of measurement - pg/mL
Mean change in albumin measured in blood | Baseline to day 15
  Unit of measurement - pg/mL
Mean change in magnesium measured in blood | Baseline to day 15
  Unit of measurement - mEq/L
Mean change in erythrocyte sedimentation rate (ESR) measured in blood | Baseline to day 15
  Unit of measurement - mm/hr
Mean change in fibroblast growth factor (FGF)-23 measured in blood | Baseline to day 15
  Unit of measurement - RU/ml
Mean change in total cholesterol measured in blood | Baseline to day 15
  Unit of measurement - mg/dl
Mean change in low density lipoprotein (LDL) measured in blood | Baseline to day 15
  Unit of measurement - mg/dl
Mean change in high density lipoprotein (HDL) measured in blood | Baseline to day 15
  Unit of measurement - mg/dl
Mean change in triglycerides measured in blood | Baseline to day 15
  Unit of measurement - mg/dl
Mean change in 8-isoprostane measured in urine | Baseline to day 15
  Unit of measurement - (ng/mg of creat)/kg
Mean change in symptoms | Baseline to day 15
  Higher scores indicate better health. Scores are transformed linearly to 0-100 range.
  The symptom list assesses the extent of bother (not at all, somewhat, moderately, very much, extremely) during the last 30 days in terms of issues particularly relevant to patients with kidney disease including soreness in muscles, pain (joint,back, chest), headaches, cramps during dialysis, bruising, itchy skin, shortness of breath, dizziness, lack of appetite, excessive thirst, numbness in hands or feet, trouble with memory, blurred vision, nausea, or other problems with the access site.
Mean change in effects of kidney disease | Baseline to day 15
  Higher scores indicate better health. Scores are transformed linearly to 0-100 range.
  Effects of kidney disease on daily life were assessed using the same five-point response scale used for the symptom/problem list and included restrictions on fluid and dietary intake, and impact on work, carrying out family responsibilities, travel, lifting objects, personal appearance, and time available to get things done.
Mean change in burden of kidney disease | Baseline to day 15
  Higher scores indicate better health. Scores are transformed linearly to 0-100 range.
  The burden of kidney disease scale assesses perceptions of frustration and interference of kidney disease in one's life using a definitely true to definitely false response scale (interferes too much with life, too much time spent dealing with it, feel frustrated dealing with it, feel like a burden on family).
Mean change in Medical Outcomes Study Short Form (MOS SF-12) physical composite | Baseline to day 15
  Higher scores indicate better health. Scores are transformed linearly to 0-100 range.
  Physical composite includes questions on how you feel about your physical health. In the survey, participants are asked if they could do things like climb stairs, move a table, or push a vacuum. How well they think they feel physically is a key measure of their health.
Mean change in Medical Outcomes Study Short Form (MOS SF-12) mental composite | Baseline to day 15
  Higher scores indicate better health. Scores are transformed linearly to 0-100 range.
  Mental composite includes questions about general health, activity limits, ability to accomplish desired tasks, depression and anxiety, energy level, and social activities.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Research Center of the University of Rochester Medical Center, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York